CLINICAL TRIAL: NCT00500461
Title: A Single-centre, Open-label, Sequential Ascending Cross Over Study to Examine Safety, Tolerability, Pharmacodynamics and Pharmacokinetics of Ascending Single Doses, Nominally 10, 30, 70 and 110µg Intravenous Doses and a Single 250µg Oral Dose of GSK233705 in Healthy Volunteers.
Brief Title: Study To Examine Safety, Tolerability And Pharmacokinetics Of Intravenous Doses And Oral Dose Of GSK233705
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AC2106213
Record Dates: First submitted 2007-07-10; First posted 2007-07-12 (Estimated); Last update posted 2017-08-07 (Actual); Status verified 2017-08

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Muscarinic Receptor Antagonist,; intravenous infusion,; pharmacokinetics; healthy subjects,; safety,; tolerability,; Anticholinergic,; oral dosing,
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Subjects receiving GSK233705 (Experimental): Each subject will receive one or more ascending doses given as a constant rate IV infusion over 30 minutes and a single oral dose of 250 microgram GSK233705 solution. IV doses will include 30, 70, 110 microgram of GSK233705 at specified time points.
  Interventions: Drug: GSK233705

INTERVENTIONS:
Drug: GSK233705 — GSK233705 will be available as IV infusion and oral solution containing Cellobiose octaacetate.

SUMMARY:
GSK233705 is being developed for the treatment of chronic obstructive pulmonary disease. This will be an open-label, dose-ascending study in 7 healthy male subjects to establish well tolerated intravenous doses and an oral dose of GSK233705. The main objective of the study is to confirm an IV and oral dose for a definitive human radiolabel metabolic study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects;
* Between the ages of 18-55 years, inclusive
* Body mass index within the range 18.0 to 30.0 kg/m2.
* Non-smokers
* Adequate venous access for intermittent cannulation
* A signed and dated written informed consent is obtained from the subject
* The subject is capable of giving informed consent
* Available to complete the study

Exclusion Criteria:

* Any clinically important abnormality identified in the following: at the screening medical assessment
* A mean QTc(B) value at screening >450msec, the QTc(B) of the 3 screening ECGs are not within 10% of the mean, a PR interval outside the range 90-210msec or an ECG that is not suitable for QT measurements
* A history of elevated resting blood pressure or a mean blood pressure higher than 140/90 mmHg at screening.
* A mean heart rate outside the range of 40-90 bpm at screening.
* History of use of tobacco- or nicotine-containing products within 6 months of screening or a positive cotinine test at screening.
* The subject has donated a unit (400ml) of blood within 60 days of screening, or, intends to donate during the study.
* The subject is currently taking regular (or course of) medication, whether prescribed or not, including herbal remedies such as St John's Wort.
* The subject has taken: prescription medications within the past 2 weeks prior to dosing, or OTC medications (except simple analgesics) within 48 hours prior to dosing, unless it is judged by the Investigator not to compromise their safety or influence the outcome of the study.
* The subject has participated in a study with a new molecular entity within a period of 3 months prior to dosing.
* The subject has tested positive for hepatitis C antibody, hepatitis B surface antigen or HIV

Ages: 25 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2007-06-04 (Actual); Primary Completion 2007-07-01 (Actual); Study Completion 2007-07-25 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of GSK233705: lead II monitoring out to 8 hours post dose, | out to 8 hours post dose
measurement of heart rate, blood pressure and ECG, Holter monitoring and laboratory data out to 24 hours and | out to 24 hours
review of adverse events ongoing through out study. | through out study.

SECONDARY OUTCOMES:
Plasma and urine concentrations of GSK233705 and derived pharmacokinetic parameters, out to 48 hours post dose. | out to 48 hours post dose.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] This study has not been published in the scientific literature.
- See also: Results for study AC2106213 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/AC2106213?search=study&search_terms=AC2106213#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: AC2106213 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: AC2106213 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: AC2106213 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: AC2106213 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: AC2106213 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: AC2106213 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: AC2106213 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register